CLINICAL TRIAL: NCT02994550
Title: Influence of FSH/LH Ratio in Controlled Ovarian Stimulation ( 2/1 Ratio vs 4/1 Ratio) in >35 Years Women Undergoing IVF
Brief Title: Influence of FSH/LH Ratio in Controlled Ovarian Stimulation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hospital de Cruces (Other)
Responsible Party: Principal Investigator, Antonia Exposito, PhD, Hospital de Cruces
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEIC E14/30
Record Dates: First submitted 2016-12-01; First posted 2016-12-16 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Sub-Fertility
Keywords: FSH; LH; IVF
MeSH Terms: conditions — Infertility | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FSH/LH 2/1 (Experimental): dose: 300IU FSHrec and 150IU LHrec
  Interventions: Drug: FSH/LH
- FSH/LH 4/1 (Experimental): dose: 300IU FSHrec and 75IU LHrec
  Interventions: Drug: FSH/LH

INTERVENTIONS:
Drug: FSH/LH

SUMMARY:
The aim of this study is to compare different FSH/LH ratios in controlled ovarian stimulation

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF cycles in Cruces University Hospital.
* Signed IVF and cryopreservation informed consent.
* Age >35 and <40 years.
* FSH levels <10 mIU/ml.

Exclusion Criteria:

* When inclusion criteria are not fulfilled

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 447 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy achievement | 3 months after drug administration
  To report our results in terms of pregnancy per embryo transfer

IPD SHARING:
Plan to Share IPD: Undecided